CLINICAL TRIAL: NCT05245201
Title: Optimizing EHR-Based Prediction Models to Improve HIV Preexposure Prophylaxis Use in Community Health Centers
Brief Title: Clinical Decision Support for PrEP
Acronym: PrEDICT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: OCHIN, Inc. (Other); Oregon Health and Science University (Other); National Institute of Mental Health (NIMH) (NIH); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PH000739A; R34MH122291 (NIH)
Record Dates: First submitted 2022-01-19; First posted 2022-02-17 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Preexposure Prophylaxis (PrEP)
Keywords: HIV; preexposure prophylaxis (PrEP); risk prediction; clinical decision support; electronic health records
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The intervention will be implemented in 2-3 clinics, with 2-3 control clinics receiving standard of care. Eligible community health centers will be those with at least 500 patients and a minimum of 10 HIV diagnoses. Clinics located in counties identified as HIV hotspots will be prioritized. Clinics specializing in HIV or sexual health care, where providers may have less need for PrEP decision support, will be excluded. Overall, 26 clinics are expected to meet these eligibility criteria, with a total of 831 incident HIV diagnoses in 2018. Of eligible clinics, 2-3 will be recruited to receive the intervention. Using a covariate-constrained matching procedure with EHR data on important covariates (e.g., urbanity and the sex, race, and age distributions of the patient population), 2-3matched control clinics will be selected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Standard of care (Active Comparator): Standard of care
  Interventions: Other: Standard of care
- Arm 2 - Clinical decision support for PrEP (Active Comparator): EHR-based decision support tools to support PrEP discussions and prescribing for patients who have increased predicted HIV risk
  Interventions: Other: Clinical decision support for PrEP

INTERVENTIONS:
Other: Standard of care — Two control clinics will be selected based on a set of matching criteria, e.g., urbanity and the sex, race, and age distributions of the patient population. Control clinics will not participate in study activities.
  Arms: Arm 1 - Standard of care
Other: Clinical decision support for PrEP — Healthcare providers at 2 intervention clinics (total of approximately 60 providers anticipated) will be prompted by an EHR-based tool to discuss PrEP with patients whose demographics and clinical history indicate increased predicted HIV risk. Providers will be offered clinical decision support tools to guide sexual health discussions and support PrEP prescribing.
  Arms: Arm 2 - Clinical decision support for PrEP

SUMMARY:
Scale-up of HIV preexposure prophylaxis (PrEP) is a key strategy of the federal initiative to end the HIV epidemic. However, healthcare providers lack tools to identify patients who are at increased risk for HIV infection and thus likely to benefit from PrEP. This pilot study will test the hypothesis that an electronic health record (EHR)-based clinical decision support system that incorporates an HIV risk prediction model can help providers identify patients at increased risk for HIV infection and improve PrEP prescribing in safety-net community health centers. The clinical decision support system will be implemented in the EHR at 2-3intervention clinics, while 2 control clinics will receive standard of care. The primary outcome is PrEP prescriptions. Other key metrics of PrEP-related care to be assessed include medication persistence, adherence to monitoring guidelines for PrEP, and rates of HIV/STI testing and diagnoses. The expected outcome is the foundation for a large-scale cluster randomized trial to test whether EHR-based clinical decision support tools for PrEP can improve PrEP prescribing and prevent new HIV infections in a national network of community health centers.

ELIGIBILITY:
Inclusion Criteria:

* Primary care providers at participating clinics who are licensed to prescribe PrEP

Exclusion Criteria:

* N/A

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
PrEP prescriptions | 9 months
  Number of patients with increased predicted HIV risk who are prescribed PrEP

SECONDARY OUTCOMES:
Feasibility of clinical decision support system | 6 months
  Rates at which providers view alerts about patients with increased predicted HIV risk and rates at which providers access the EHR-based decision support tools using Epic date-time stamps
Acceptability of clinical decision support system | 6 months
  One-on-one feedback interviews with clinic administrators and 3-5 providers at intervention clinics

CONTACTS AND LOCATIONS:
Overall Officials: Julia Marcus, PhD, Principal Investigator — Harvard Pilgrim Health Care Institute; Douglas Krakower, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Saban Community Clinic, Los Angeles, California
  - Roanoke Chowan Community Health Center, Ahoskie, North Carolina
  - Kintegra Health, Gastonia, North Carolina

IPD SHARING:
Plan to Share IPD: No